CLINICAL TRIAL: NCT02509351
Title: Randomized, Placebo-controlled Double Blind Study of Preoperative Misorostol for Reduction of Intraoperative Bleeding in Women Delivered by Ceserean Section
Brief Title: Could Pre-operative Rectal Misoprostol Reduce Intra-operative Blood Loss During Ceserean Section?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POMCS
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-05

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol (Experimental): women receiving pre-operative rectally administered 400 microgram misoprostol
  Interventions: Drug: misoprostol
- placeboo (Active Comparator): women receiving placebo
  Interventions: Drug: placeboo

INTERVENTIONS:
Drug: misoprostol — 400 microgram of misoprostol is given preoperatively in patients undergoing elective cesarean section
  Other Names: mesotac
  Arms: misoprostol
Drug: placeboo — women will recive 2 identical tablets as placeboo
  Other Names: control
  Arms: placeboo

SUMMARY:
* Misoprostol reduces the uterine bleeding after cesarean delivery without harmful effects on either mother or baby.
* The aim of the this study is to address if there is any benefits 'regarding the intra-operative blood loss' from preoperative rectal administration of 400 mic of Misoprostol in addition to the routinely administrated 10 units of oxytocin

DETAILED DESCRIPTION:
Research question:

In women undergoing elective ceserean section, is preoperative 400 mic Misoprostol reduce intra-operative blood loss?

Research hypothesis:

pre-operative Misoprostol doesn't reduce intraoperative blood loss in women undergoing ceserean section

ELIGIBILITY:
Inclusion Criteria:

* 38-41 weeks of amenorrhea
* scheduled for elective lower segment cesarean section

Exclusion Criteria:

* confirmed intrauterine fetal death
* more than previous 2 ceserean sections
* multiple pregnancy
* antepartum haemorrhage
* self-reported maternal heart disease
* current diagnosis of severe malaria or acute bacterial infection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
volume of intraoperative blood loss | 30 minute
  volume of intraoperative blood loss will be measured in "cc" by a didcated nurse who will use separate suction sets to differentiate between blood and liquor

SECONDARY OUTCOMES:
maternal mortality | 6 months
mean measured blood loss | 1, 2, and 24 h postpartum
placental retention | 30 minutes
  when the placenta is not delivered spontaneously for 30 minutes
requirement for blood transfusion | 24 hours
  indicated per clinical protocol at the study site for mothers with a hemoglobin <100 g/l and/or severe pallor
requirement for additional management of PPH, including therapeutic uterotonic drugs or surgical or radiological procedures | 24 hours
postpartum hemoglobin | 24 hours
  less than 10gm%
mean postpartum hematocrit | 24 hours
  more than 10% drop in the postpartum hematocrit

CONTACTS AND LOCATIONS:
Overall Officials: Helmy Dr metawe, MD, Study Chair — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No